CLINICAL TRIAL: NCT03609853
Title: Behavioral Pharmacology of THC and D-limonene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00085652; R01DA043475 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: D-limonene and THC Pharmacodynamics
MeSH Terms: interventions — Limonene; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Placebo (Placebo Comparator): Placebo (5mL distilled water)
  Interventions: Drug: Placebo
- Vaporized low THC (Experimental): 15mg of pure THC
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- Vaporized high THC (Experimental): 30mg of pure THC
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- Vaporized low d-limonene (Experimental): 1mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- Vaporized high d-limonene (Experimental): 5mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- Low THC and low d-limonene (Experimental): 15mg of THC paired with 1mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- High THC and low d-limonene (Experimental): 30mg of THC paired with 1mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- Low THC and high d-limonene (Experimental): 15mg of THC paired with 5mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- High THC and high d-limonene (Experimental): 30mg of THC paired with 5mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene
- High THC and 15mg d-limonene (Experimental): 30mg of THC paired with 15mg of d-limonene
  Interventions: Drug: Vaporized THC, limonene, or THC and limonene

INTERVENTIONS:
Drug: Placebo — Placebo vapor (distilled water)
  Arms: Placebo
Drug: Vaporized THC, limonene, or THC and limonene — Acute drug exposure
  Arms: High THC and 15mg d-limonene; High THC and high d-limonene; High THC and low d-limonene; Low THC and high d-limonene; Low THC and low d-limonene; Vaporized high THC; Vaporized high d-limonene; Vaporized low THC; Vaporized low d-limonene

SUMMARY:
This study will evaluate the pharmacokinetics and pharmacodynamics of vaporized d-limonene and THC administered via inhalation.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). Participants will complete 9 acute drug administration periods in which they will administer THC alone, limonene alone, THC and limonene together, or placebo. Subjective drug effects and vital signs will be assessed following drug administration. Each participant will receive all 9 dose conditions in a randomized order using a placebo controlled within-subject crossover design. The study will help us understand the individual and interactive effects of THC and d-limonene, two common constituents found in cannabis.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
4. Test negative for drugs of abuse other than cannabis, including breath alcohol at the screening visit and at clinic admission
5. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
6. Have a body mass index (BMI) in the range of 18 to 36 kg/m2
7. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
8. Have no allergies to any of the ingredients used to prepare vapor (THC, d-limonene).
9. Report having experienced anxiety after consuming cannabis in the past.

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
2. History of or current evidence of significant medical (e.g. seizure disorder) or psychiatric illness (e.g. psychosis) judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an over the counter, systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
5. Use of dronabinol (Marinol®) within the past month.
6. Average use of cannabis more than 2 times per week in the prior 3 months.
7. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
8. Abnormal EKG result that in the investigator's opinion is clinically significant.
9. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
10. Having previously sought medical attention to manage adverse effects following acute cannabis use.
11. Individuals with anemia or who have donated blood in the prior 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a within-subjects design, so all participants were exposed to all 10 conditions in a randomized order.
Groups:
- Vaporized Delta-9-tetrahydrocannabinol (THC) With and Without Limonene: Participants vaporized THC and limonene in a within-subject crossover design:
  1. Placebo
  2. Low THC (15mg)
  3. High THC (30mg)
  4. Low Limonene (1mg)
  5. High Limonene (5mg)
  6. Low THC (15mg) + low Limonene (1mg)
  7. High THC (30mg) + low Limonene (1mg)
  8. Low THC (15mg) + high Limonene (5mg)
  9. High THC (30mg) + high Limonene (5mg)
  10. High THC (30mg) + 15mg Limonene
Period: Overall Study
Arm/Group | Vaporized Delta-9-tetrahydrocannabinol (THC) With and Without Limonene
Started | 35
Placebo | 28
Vaporized Low Delta-9-tetrahydrocannabinol (THC) | 25
Vaporized High THC | 27
Vaporized Low D-limonene | 30
Vaporized High D-limonene | 27
Low THC and Low D-limonene | 27
High THC and Low D-limonene | 31
Low THC and High D-limonene | 25
High THC and High D-limonene | 26
High THC and 15mg Limonene | 12
Completed | 20
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: We are reporting data for study completers. 20 participants completed the study.
Groups:
- Vaporized THC With and Without Limonene: All study completers completed the following 10 conditions in a randomized order:
  1. Placebo (distilled water)
  2. Vaporized Low THC (15mg)
  3. Vaporized High THC (30mg)
  4. Vaporized Low d-Limonene (1mg)
  5. Vaporized High d-Limonene (5mg)
  6. Vaporized Low THC + low d-Limonene
  7. Vaporized High THC + low d-Limonene
  8. Vaporized Low THC + high d-Limonene
  9. Vaporized High THC + high d-Limonene
  10. Vaporized High THC + 15mg d-Limonene
Arm/Group | Vaporized THC With and Without Limonene
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 26 [20 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Change From Baseline Anxiety as Assessed by the Drug Effect Questionnaire (DEQ)
Description: Peak rating (0-100) of Anxiety on the DEQ, a visual analog scale (VAS) self-report questionnaire with 0 being No anxiety and 100 being maximum anxiety
Time Frame: 0-6 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaporized Low THC | Vaporized High THC | Vaporized Low D-limonene | Vaporized High D-limonene | Low THC and Low D-limonene | High THC and Low D-limonene | Low THC and High D-limonene | High THC and High D-limonene | High THC and 15mg D-limonene
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 12
score on a scale | -1.2 (8.1) | 13.8 (26.5) | 18.7 (25.7) | -1.9 (13.9) | -0.9 (6.8) | 8.7 (26) | 19.5 (22.1) | 10.2 (14.9) | 14 (21.5) | 4.3 (21.9)

2. Secondary Outcome: Mean Peak Change From Baseline Paranoid as Assessed by the Drug Effect Questionnaire (DEQ)
Description: Peak change from baseline rating of Paranoid on the DEQ, a 100pt VAS scale with 0 being no paranoia and 100 being extreme paranoia
Time Frame: 0-6 hours
Population: Study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaporized Low THC | Vaporized High THC | Vaporized Low D-limonene | Vaporized High D-limonene | Low THC and Low D-limonene | High THC and Low D-limonene | Low THC and High D-limonene | High THC and High D-limonene | High THC and 15mg D-limonene
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 12
score on a scale | -0.4 (1.6) | 11.1 (21.7) | 14.6 (22.2) | 1.3 (4.8) | -0.6 (2.9) | 9.9 (17.8) | 16.1 (23.4) | 9.3 (19.1) | 7.3 (14.8) | 6.3 (16.9)

3. Secondary Outcome: Mean Peak Change From Baseline Subjective "Heart Racing" as Assessed by the Drug Effect Questionnaire (DEQ)
Description: Mean peak change from baseline for subjective heart racing on the DEQ, a 0-100 VAS scale with 0 being no feeling of heart racing and 100 being an extreme feeling of heart racing.
Time Frame: 0-6 hours
Population: Study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaporized Low THC | Vaporized High THC | Vaporized Low D-limonene | Vaporized High D-limonene | Low THC and Low D-limonene | High THC and Low D-limonene | Low THC and High D-limonene | High THC and High D-limonene | High THC and 15mg D-limonene
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 12
score on a scale | 0.1 (3.1) | 25.2 (28.7) | 32.5 (25.7) | 4.3 (12.1) | 1.1 (9.6) | 21.2 (28.7) | 34 (26.1) | 16.8 (21.8) | 23.2 (21.1) | 24.5 (25.8)

4. Secondary Outcome: Mean Peak Change From Baseline Heart Rate
Description: Peak change from baseline in Heart Rate (bpm) measured in seated position by automated monitor
Time Frame: 0-6 hours
Population: Study completers
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Vaporized Low THC | Vaporized High THC | Vaporized Low D-limonene | Vaporized High D-limonene | Low THC and Low D-limonene | High THC and Low D-limonene | Low THC and High D-limonene | High THC and High D-limonene | High THC and 15mg D-limonene
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 12
Beats per minute | 0.8 (17.6) | 17 (21) | 24.8 (23.1) | -0.4 (12.7) | -1.1 (13.7) | 19.5 (25.3) | 24.1 (24.7) | 19.6 (19.9) | 28.5 (9.5) | 27.8 (14.2)

ADVERSE EVENTS:
Time Frame: 0-6 hours
Description: International Council for Harmonisation (ICH) guidelines are followed for Adverse Event (AE) reporting, as AEs occur they are documented.
Arm/Group | Placebo | Vaporized Low THC | Vaporized High THC | Vaporized Low D-limonene | Vaporized High D-limonene | Low THC and Low D-limonene | High THC and Low D-limonene | Low THC and High D-limonene | High THC and High D-limonene | High THC and 15mg D-limonene
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25 | 0/27 | 0/30 | 0/27 | 0/27 | 0/31 | 0/25 | 0/26 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/27 | 0/30 | 0/27 | 0/27 | 0/31 | 0/25 | 0/26 | 0/12
Other Adverse Events (participants affected / at risk) | 0/28 | 1/25 | 3/27 | 2/30 | 0/27 | 3/27 | 4/31 | 0/25 | 2/26 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Vaporized Low THC (N=25) | Vaporized High THC (N=27) | Vaporized Low D-limonene (N=30) | Vaporized High D-limonene (N=27) | Low THC and Low D-limonene (N=27) | High THC and Low D-limonene (N=31) | Low THC and High D-limonene (N=25) | High THC and High D-limonene (N=26) | High THC and 15mg D-limonene (N=12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intrusive Anxiety (Social circumstances) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Anxiety that interfered with functioning and caused discomfort to the point that participant reported it to medical staff
Lightheaded (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Heart Rate of >120 Beats Per Minute

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03609853/Prot_000.pdf